CLINICAL TRIAL: NCT04194593
Title: Development of a New Algorithm-based Classification for Glioma
Brief Title: Biomarker-based Algorithm for Diagnosis of Glioma
Acronym: TELOGNOSTIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0795
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glioma: FFPE (Formalin-Fixed Paraffin-Embedded) or frozen samples will be used for DNA extraction. Different gliomas tumors will be used (oligodendroglioma, astrocytomas, glioblastoma)
  Interventions: Other: PCR (Polymerase Chain Reaction)

INTERVENTIONS:
Other: PCR (Polymerase Chain Reaction) — Biological testing of FFPE (Formalin-Fixed Paraffin-Embedded) or frozen samples of tumors will be led. These tissues have been collected during the treatment of patients (for diagnostic purposes).
  A molecular analysis (polymerase chain reaction) is led on DNA extracted from FFPE/frozen conserved tissues, and a result is produced by the algorithm.

SUMMARY:
ATRX (X-linked mental retardation and alpha-thalassaemia syndrome protein) loss and pTERT (Telomerase reverse transcriptase) mutation are diagnostic markers of gliomas. However, 4 to 28% of gliomas shows none of these alterations. The aim of this project is to propose a new test able to detect the telomeric status for every glioma. Based on this test and other markers (such as mutation of IDH1 (isocitrate dehydrogenase 1) and IDH2 (isocitrate dehydrogenase 2)), investigators propose an algorithm, able to classify the main subtypes of gliomas (astrocytoma, oligodendroglioma and glioblastoma).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of glioma (retrospective),
* Patient with available biological material : extracted DNA and/or FFPE tissue and/or frozen sample.
* Samples are not required any more for diagnosis purpose
* Patient with informed consent

Exclusion Criteria:

* Patient with no informed consent
* Patients with no available biological sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 samples of gliomas (FFPE and/or frozen tissues)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the prognosis and diagnosis values of a new qPCR (quantitative polymerase chain reaction) -based biological testing in glioma | 1 year
  An algorithm will be built, based on the result of this specific biological testing combined with other markers (determined in routine clinical testing). The algorithm parameters will be set using samples with a clear diagnosis (concordant molecular and immuno-histological markers). Then gliomas with uncertain diagnosis will be classified and the global overall survival will be predicted.
  Biological testing will be performed during one year and the analyses in terms of disease outcome will be refreshed every year.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Pathologie Est, Biopathologie moléculaire, Hôpitaux Est, HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No